CLINICAL TRIAL: NCT06647277
Title: An Open-Label Phase I Clinical Trial of Vancomycin Followed by Fecal Microbiota Transplant for the Treatment of Parkinson's Disease
Brief Title: Fecal MicrobiotaTransplant for the Treatment of Parkinson's Disease
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ProgenaBiome (Other)
Responsible Party: Principal Investigator, Sabine Hazan, Principal Investigator, ProgenaBiome
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRG-056
Record Dates: First submitted 2024-10-08; First posted 2024-10-17 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Fecal Microbiota Transplantation; Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- PD patients (Other): This is an open-label clinical trial to evaluate the Safety of fecal microbiota transplant following a 10 day treatment with Vancomycin in adult subjects with Parkinson's disease.
  Interventions: Combination Product: Fecal Microbiota Transplant

INTERVENTIONS:
Combination Product: Fecal Microbiota Transplant — Fecal Microbiota Transplant
  Other Names: Vancomycin

SUMMARY:
FMT may significantly improve quality of life and Parkinson Disease (PD) symptom severity measurements. We hypothesize that gut microbial dysbiosis is a major contributing factor in Parkinson's disease.

DETAILED DESCRIPTION:
This is an open-label clinical trial to evaluate the Safety of fecal microbiota transplant following a 10 day treatment with Vancomycin in adult subjects with Parkinson's disease. Subjects in the study are required to meet with the study clinician on 11 occasions: two (2) visits for informed consent and baseline assessment, one (1) visit prior to FMT for colonoscopy instructions and exam, one (1) visit for the fecal microbiota transplant procedure by colonoscopy at an outpatient surgical center, seven (7) visits for post-FMT assessment. There are also daily phone calls in the week following the FMT, and weekly phone call visits (during weeks in which there is not a physical visit) to check up on how the subject is doing, any change in medications, side effects, and answer any questions.

ELIGIBILITY:
Inclusion Criteria:

* Individuals diagnosed with PD

Exclusion Criteria:

* Non-PD individuals

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Parkinson's disease symptoms | 6.5 months for each subject
  Changes in symptoms reported

SECONDARY OUTCOMES:
Alterations in Subject microbiome from baseline | 6.5 months for each subject
  Changes in microbiome Shannon Diversity Index and relative abundance

CONTACTS AND LOCATIONS:
Locations (1):
- Sabine Hazan, Ventura, California, United States

IPD SHARING:
Plan to Share IPD: No